CLINICAL TRIAL: NCT02639728
Title: Prospective Study of the Effect of Coffee Consumption in Enhancing Recovery of Bowel Function Following Colorectal Surgery.
Brief Title: The Effect of Coffee Consumption in Enhancing Recovery of Bowel Function Following Colorectal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yosef Nasseri, MD, MD, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030891
Record Dates: First submitted 2015-12-10; First posted 2015-12-24 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Ileus
Keywords: Bowel surgery; Postoperative bowel recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regular coffee (Experimental): Will receive a 4oz cup coffee, three times daily (at 8:00, 12:00, and 16:00 hours)and instructed to consume the entirety of its liquid contents. This liquid consumption will begin on the morning of POD #1 at 8:00 hours. Duration of experimental treatment will last until first flatus or bowel movement or 7 days, whichever comes first.
  Interventions: Other: Regular Coffee
- Decaffeinated coffee (Experimental): Will receive a 4oz cup of decaffeinated coffee (at 8:00, 12:00, and 16:00 hours) and instructed to consume the entirety of its liquid contents. This liquid consumption will begin on the morning of POD #1 at 8:00 hours. Duration of experimental treatment will last until first flatus or bowel movement or 7 days, whichever comes first.
  Interventions: Other: Decaffeinated coffee
- Warm water (Experimental): Will receive a 4oz cup of warm water at 8:00, 12:00, and 16:00 hours) and instructed to consume the entirety of its liquid contents. This liquid consumption will begin on the morning of POD #1 at 8:00 hours. Duration of experimental treatment will last until first flatus or bowel movement or 7 days, whichever comes first.
  Interventions: Other: Warm water

INTERVENTIONS:
Other: Regular Coffee — Regular coffee will be given a 4oz cup three times daily and will be instructed to consume all of its liquid contents.
  Arms: Regular coffee
Other: Decaffeinated coffee — Decaffeinated coffee will be given a 4oz cup three times daily and will be instructed to consume all of its liquid contents.
  Arms: Decaffeinated coffee
Other: Warm water — Warm water will be given a 4oz cup three times daily and will be instructed to consume all of its liquid contents.
  Arms: Warm water

SUMMARY:
The effects of coffee have been shown to act as a colonic stimulant. Caffeinated coffee stimulates colonic activity, most notably in the transverse/descending colon, in magnitude similar to a meal, 60% stronger than water, and 23% stronger than decaffeinated coffee. [1] Moreover, the consumption of both water and caffeine causes a decrease in the rectal sensory threshold for the desire to defecate, while anal sphincter pressure after caffeine intake is significantly higher than after water intake. This may result in an earlier desire to defecate. [2] Coffee has also been shown to have an effect on defecation by increasing rectal tone by 45% (measured with a barostat) thirty minutes after consumption. [3]

DETAILED DESCRIPTION:
Study Objectives

Primary objective: To determine if the use of coffee in the postoperative period will reduce time to recovery of GI function by at least one day in patients undergoing elective colorectal operations. (This will be assessed by twice daily interview of patients as to whether they have passed flatus or had a bowel movement)

Secondary objective: To determine if the use of coffee in the postoperative period will reduce hospital length of stay by at least one day, and to also evaluate the tolerance of solid food, which will help determine postoperative ileus and rates of vomiting/nasogastric tube (re)insertion, and other perioperative morbidities such as anastomotic leak, wound infection, and intra-abdominal abscesses in patients undergoing elective colorectal operations.

Study Design

This study involves the evaluation of patients who consume coffee compared with patients who consume warm water during the postoperative period after elective colorectal surgery with primary anastomosis.

This study will be a single-center, randomized trial. Patients who undergo elective colorectal surgery at Cedars-Sinai Medical Center and agree to participate in the study will be randomized 1:1:1 to those who drink regular coffee, decaffeinated coffee, and no coffee. Randomization will occur via an online program (www.randomizer.org), which assigns participants to experimental conditions. The subjects assigned to drink regular coffee, decaffeinated coffee, or warm water will be given a 4oz cup three times daily and will be instructed to consume all of its liquid contents.

Postoperative care will otherwise be the same for all subjects, as dictated by the clinical judgment of the surgical team.

ELIGIBILITY:
Inclusion Criteria:

* • Patients due to undergo small and/or large partial bowel resection via laparotomy or laparoscopy with primary anastomosis. Planned postoperative care includes removing the NG tube at the end of surgery and clear liquid diet of POD #1.

  * Patients, both male and female, must be between the ages of 18-85.
  * Patients must be able to freely give written informed consent to participate in the study and have signed the Informed Consent Form.

Exclusion Criteria:

* • Study patients who do not meet inclusion criteria will not qualify for study inclusion.

  * Patients with a history of prior intestinal surgery, excluding appendectomy.
  * Patients who require an ostomy during their elective colorectal surgery.
  * Patients who require postoperative ventilation, pressors, or ICU stay.
  * Those who are mentally incompetent, unable, or unwilling to provide informed consent or comply with study procedures.
  * American Society of Anesthesiologist (ASA) class IV or V.
  * Those with a history of carcinomatosis.
  * Those with a history of radiation enteritis.
  * Women who are pregnant.
  * Patients who have a history of epilepsy.
  * Patients with prior cardiovascular disorders including uncontrolled hypertension, prior myocardial infarction, or heart failure.
  * Patients with peptic ulcers.
  * Patients with glaucoma.
  * Non-English Speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
GI Function | 30 days
  Time to first flatus and/or bowel movement as assessed twice per day by inquiry from the primary team and study investigators.

SECONDARY OUTCOMES:
Hospital Days | 30 days
  Evaluation of length of postoperative hospital stay, will be recorded from medical records.
Vomiting | 30 days
  Evaluation of number of episodes of vomiting will be collected from medical records
Nasogastric tube | 30 days
  Number of nasogastric tube (re)insertion, will be collected from medical records
Anastomotic leak | 30 days
  Evaluation of any anastomotic leak will be collected from medical records
Wound Infection | 30 days
  Evaluation for any wound infection will be collected from medical records
Abscesses | 30 days
  Evaluation for any intra-abdominal abscess will be collected from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Nasseri, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Yosef Nasseri, MD, Los Angeles, California, United States

REFERENCES:
- [Background] Rao SS, Welcher K, Zimmerman B, Stumbo P. Is coffee a colonic stimulant? Eur J Gastroenterol Hepatol. 1998 Feb;10(2):113-8. doi: 10.1097/00042737-199802000-00003. PMID 9581985
- [Background] Lohsiriwat S, Kongmuang P, Leelakusolvong S. Effects of caffeine on anorectal manometric findings. Dis Colon Rectum. 2008 Jun;51(6):928-31. doi: 10.1007/s10350-008-9271-y. Epub 2008 Mar 19. PMID 18350336
- [Background] Sloots CE, Felt-Bersma RJ, West RL, Kuipers EJ. Stimulation of defecation: effects of coffee use and nicotine on rectal tone and visceral sensitivity. Scand J Gastroenterol. 2005 Jul;40(7):808-13. doi: 10.1080/00365520510015872. PMID 16109656
- [Background] Muller SA, Rahbari NN, Schneider F, Warschkow R, Simon T, von Frankenberg M, Bork U, Weitz J, Schmied BM, Buchler MW. Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy. Br J Surg. 2012 Nov;99(11):1530-8. doi: 10.1002/bjs.8885. Epub 2012 Sep 14. PMID 22987303
- [Derived] Nasseri Y, Kasheri E, Oka K, Zhu R, Smiley A, Cohen J, Ellenhorn J, Barnajian M. Does coffee affect bowel recovery following minimally invasive colorectal operations? A three-armed randomized controlled trial. Int J Colorectal Dis. 2023 Jul 20;38(1):199. doi: 10.1007/s00384-023-04494-7. PMID 37470901